CLINICAL TRIAL: NCT03754569
Title: Microscopic Peritoneal Metastases After Complete Macroscopic Cytoreductive Surgery for Epithelial Ovarian Cancer
Acronym: MicroPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K171203J
Record Dates: First submitted 2018-07-16; First posted 2018-11-27 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-01

CONDITIONS: Epithelial Ovarian Cancer
Keywords: ovarian; peritoneal; recurrences; surgery; cancer; metastases
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Recurrence; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peritoneal biopsies (Experimental): We will perform at the end of complete macroscopic cytoreductive surgery (CC-0) for epithelial ovarian cancer random peritoneal biopsies in apparently healthy peritoneum in order to assess the presence of microscopic peritoneal metastases
  Interventions: Procedure: Peritoneal biopsies after complete macroscopic cytoreduction

INTERVENTIONS:
Procedure: Peritoneal biopsies after complete macroscopic cytoreduction — We will perform at the end of complete macroscopic cytoreductive surgery (CC-0) for epithelial ovarian cancer random peritoneal biopsies in apparently healthy peritoneum in order to assess the presence of microscopic peritoneal metastases

SUMMARY:
The objective of the cytoreductive surgery carried out for the management of ovarian cancers is to obtain a complete macroscopic cytoreduction. This means that all visible peritoneal metastases must be resected. The peritoneum is the most frequent site of recurrence after initial management. There is no data on the existence, prevalence of microscopic peritoneal metastases. It nevertheless represents a therapeutic target (intraperitoneal chemotherapy). The main objective is the demonstration of microscopic peritoneal metastases in macroscopically healthy peritoneum after complete macroscopic cytoreductive surgery.

DETAILED DESCRIPTION:
Understanding biology and progression mechanisms of peritoneal metastases (PM) of epithelial ovarian cancer (EOC) is a cornerstone in the knowledge and the comprehensive management of the disease, as PM will occur in the majority of patients. Indeed, the goal of cytoreductive surgery (CRS) in these patients is to completely remove all visible peritoneal invasion because the absence of residual disease after surgery is known to improve the prognosis.

Despite clinical remission after the completion of complete surgery and platinum-based chemotherapy, 60% of patient develop peritoneal recurrence. This suggests that microscopic lesions may be present that are not eradicated by surgery, not controlled by systemic chemotherapy and that may be one of the mechanisms leading to peritoneal recurrence. Peritoneal carcinomatosis is responsible for the greatest morbidity and mortality in women with EOC.

There are very few studies in the literature on microscopic peritoneal involvement in EOC, its detection and potential role in the progression of cancer. The peritoneum should be considered an organ in its own right and the surgeon must treat peritoneal metastases with the intent to cure. To follow the recommendations, this microscopic disease must be managed, because complete CRS is now a skill that can be mastered skill and its uses is a validated guideline. Moreover, "complete CRS" should be defined as "without macroscopic residual disease" thus highlighting the presence of microscopic disease.

The goal of this study is to add scientific evidence for the existence of Microscopic Peritoneal Metastases (mPM) and to justify the need for additional diagnostic and therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old, French nationality
* with epithelial ovarian or tubal cancer
* Complete macroscopic cytoreductive surgery (CC-0) regardless of the sequence compared to chemotherapy.
* Patient giving express consent

Exclusion Criteria:

* Borderline ovarian tumor
* Incomplete cytoreductive surgery
* Pregnant women
* Major under guardianship / trusteeship,
* Not insured

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Identification of microscopic peritoneal metastases on pathological examination of peritoneal biopsies after complete macroscopic cytoreductive surgery for epithelial ovarian cancer. | one year
  Random peritoneal biopsies in apparently healthy peritoneum, will be performed at the end of complete macroscopic cytoreductive surgery (CC-0) for epithelial ovarian cancer. If peritoneal metastases are identified on this sample, they will be the subject of a detailed morphological description.
  Presence of microscopic peritoneal metastases will be measured (µm) using light microscope on HE slides from formalin fixed paraffin embedded tissues, by two different expert pathologists

SECONDARY OUTCOMES:
Expression of folate receptor by microscopic peritoneal metastases and comparison with primary tumor | one year
  Expression of folate receptor will measured by immuno-histo-chemistry. The intensity of the expression will be evaluated using semiquantitative method.
  Expression of folate receptor by microscopic peritoneal metastases will be assessed using immunohistochemistry with mouse monoclonal NCL-L-FRalpha antibody (Leica Biosystems). Expression will be quantified with a light microscope, using H-score according to the following formula : H-score = [1 × (% cells 1+) + 2 × (% cells 2+) + 3 × (% cells 3+)].

CONTACTS AND LOCATIONS:
Overall Officials: Henri M AZAIS, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided